CLINICAL TRIAL: NCT05226598
Title: A Randomized, Double-Blind, Phase 3 Study of Pembrolizumab/Vibostolimab Coformulation (MK-7684A) in Combination With Chemotherapy Versus Pembrolizumab Plus Chemotherapy as First Line Treatment for Participants With Metastatic Non-Small Cell Lung Cancer (MK-7684A-007/KEYVIBE-007)
Brief Title: Study of Pembrolizumab/Vibostolimab Coformulation (MK-7684A) in Combination With Chemotherapy Versus Pembrolizumab Plus Chemotherapy in Participants With Metastatic Non-Small Cell Lung Cancer (MK-7684A-007/KEYVIBE-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7684A-007; MK-7684A-007 (Other: MSD); KEYVIBE-007 (Other: MSD); jRCT2031220098 (Registry Identifier: jRCT); 2023-506074-12-00 (Registry Identifier: EU CT); U1111-1293-2114 (Registry Identifier: UTN)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Cisplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-7684A + Chemotherapy (Experimental): Participants receive pembrolizumab/vibostolimab (co-formulation of 200mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 35 cycles (up to ~2 years) PLUS paclitaxel IV (on Day 1 of each cycle) OR nab-paclitaxel IV (on Days 1, 8, and 15 of each cycle) and carboplatin IV (on Day 1 of each cycle) for 4 cycles for Squamous NSCLC; PLUS carboplatin IV (on Day 1 of each cycle) Or cisplatin IV (on Day 1 of each cycle) for 4 cycles and pemetrexed IV (on Day 1 of each cycle) until progression, intolerable adverse events, or participant/physician decision for Non-squamous.
  Interventions: Biological: Pembrolizumab/Vibostolimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Pemetrexed
- Pembrolizumab + Chemotherapy (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 35 cycles (up to ~2 years) PLUS paclitaxel IV (on Day 1 of each cycle) OR nab-paclitaxel IV (on Days 1, 8, and 15 of each cycle) and carboplatin IV (on Day 1 of each cycle) for 4 cycles for Squamous NSCLC; PLUS carboplatin IV (on Day 1 of each cycle) Or cisplatin IV (on Day 1 of each cycle) for 4 cycles and pemetrexed IV (on Day 1 of each cycle) until progression, intolerable adverse events, or participant/physician decision for Non-squamous.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Pemetrexed; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab/Vibostolimab — Co-formulation of pembrolizumab 200 mg/20 mL vial and vibostolimab 200 mg administered as IV infusion for up to 35 administrations
  Other Names: MK-7684A
  Arms: MK-7684A + Chemotherapy
Drug: Carboplatin — Carboplatin 10 mg/ml administered as IV infusion Q3W for 4 administrations
  Other Names: PARAPLATIN®, Paraplatin NovaPlus ®
Drug: Cisplatin — Cisplatin 1 mg/ml administered as IV infusion Q3W for 4 administrations
  Other Names: Platinol-AQ®
Drug: Paclitaxel — Paclitaxel 6mg/ml administered as IV infusion Q3W for 4 administrations
  Other Names: TAXOL®, ONXOL®
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/vial administered as IV infusion Days 1, 8, and 15 of each 21-day cycle for 4 administrations
  Other Names: ABRAXANE®
Drug: Pemetrexed — Pemetrexed 500 mg/vial administered as IV infusion Q3W until progression, intolerable adverse event (AE), or participant or physician decision
  Other Names: Alimta®
Biological: Pembrolizumab — Pembrolizumab 25 mg/mL administered as IV infusion Q3W for up to 35 administrations
  Other Names: MK-3475, KEYTRUDA®
  Arms: Pembrolizumab + Chemotherapy

SUMMARY:
The primary hypothesis is that pembrolizumab/vibostolimab (MK-7684A) in combination with chemotherapy is superior to pembrolizumab in combination with chemotherapy with respect to overall survival (OS) in participants with programmed cell death-ligand 1 (PD-L1) tumor proportion score (TPS) ≥1%.

DETAILED DESCRIPTION:
Effective as of Amendment 5, Participants receiving coformulation of pembrolizumab/vibostolimab plus chemotherapy will be transitioned to standard of care (SOC, pembrolizumab plus chemotherapy). Participants with access to approved standard of care (SOC) should be considered for discontinuation from the study. Those benefiting from pembrolizumab plus chemotherapy, but unable to access it as SOC outside the study, may continue on study and receive treatment with pembrolizumab plus chemotherapy until discontinuation criteria are met.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* A histologically or cytologically confirmed diagnosis of Stage IV squamous or non-squamous NSCLC
* Has not received prior systemic treatment for metastatic NSCLC
* Has measurable disease based on RECIST 1.1, as determined by the local site assessment
* Has a life expectancy of at least 3 months
* Males: Use contraception unless confirmed to be azoospermic; Females: Women of childbearing potential use highly effective contraceptive method

Exclusion Criteria:

* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Severe hypersensitivity to MK-7684, MK-7684A, pembrolizumab, chemotherapy components, and/or any of its excipients
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study medication
* Active autoimmune disease that has required systemic treatment in past 2 years, except replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid)
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV), Hepatitis B or/and Hepatitis C virus
* Received prior systemic anticancer therapy for metastatic disease
* Received a live or live attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed
* History of allogeneic tissue/solid organ transplant
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g/day, for a 5-day period (8-day period for long-acting agents, such as piroxicam)
* Is unable or unwilling to take folic acid or vitamin B12 supplementation
* Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2026-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (149):
- United States (12):
  - UCHealth Memorial Hospital-Heme Onc ( Site 0003), Colorado Springs, Colorado
  - University of Colorado Health - Harmony-Cancer Care and Hematology - Ft. Collins ( Site 0031), Fort Collins, Colorado
  - Mayo Clinic in Florida ( Site 0022), Jacksonville, Florida
  - Mount Sinai Hospital ( Site 0011), Chicago, Illinois
  - University of Chicago Medical Center ( Site 0015), Chicago, Illinois
  - New England Cancer Specialists ( Site 0008), Scarborough, Maine
  - Cancer and Hematology Centers of Western Michigan ( Site 0002), Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Minnesota ( Site 0030), Rochester, Minnesota
  - Stony Brook University-Cancer Center ( Site 0013), Stony Brook, New York
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute ( Site 0012), Lancaster, Pennsylvania
  - Charleston Oncology ( Site 0019), Charleston, South Carolina
  - University of Virginia Cancer Center ( Site 0018), Charlottesville, Virginia
- Argentina (7):
  - Centro de Oncología e Investigación de Buenos Aires ( Site 0203), Berazategui, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0204), Mar del Plata, Buenos Aires
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 0209), ABB, Buenos Aires F.D.
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC)-Medical Oncology ( Site 0202), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 0205), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 0212), Rosario, Santa Fe Province
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0206), La Rioja
- Austria (6):
  - Medizinische Universität Graz ( Site 0704), Graz, Styria
  - Medizinische Universitaet Innsbruck ( Site 0703), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen-Department of Pneumology ( Site 0705), Linz, Upper Austria
  - Kepler Universitätsklinikum ( Site 0707), Linz, Upper Austria
  - Klinik Penzing-2. Lungenabteilung ( Site 0702), Vienna, Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 0701), Vienna
- Brazil (5):
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0403), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0405), Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia Reichow ( Site 0407), Blumenau, Santa Catarina
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA ( Site 0406), Rio de Janeiro
  - Hospital Paulistano ( Site 0401), São Paulo
- Chile (8):
  - FALP-UIDO ( Site 0505), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión ( Site 0515), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0510), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 0502), Temuco, Región de la Araucanía
  - CIDO SpA-Oncology ( Site 0508), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0503), Viña del Mar, Región de Valparaíso
  - Biocenter ( Site 0514), Concepción, Región del Biobío
  - Centro de Investigación Oncológica del Norte ( Site 0504), Antofagasta
- China (28):
  - Anhui Provincil Hospital South District-Respiratory Medicine Dept ( Site 2619), Hefei, Anhui
  - Beijing Cancer hospital-Thoracic Cancer Department A ( Site 2602), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital-oncology department ( Site 2621), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 2626), Xiamen, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine (, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital-oncology of department ( Site 2604), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2608), Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 2618), Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 2617), Wuhan, Hubei
  - Xiangya Hospital Central South University-Oncology department ( Site 2627), Changsha, Hunan
  - The Second Xiangya Hospital of Central South University ( Site 2623), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 2622), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Oncology (, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University-Respiratory Medicine Department ( Site 2625), Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University-Oncology Department ( Site 2624), Nanchang, Jiangxi
  - Jilin Cancer Hospital-oncology department ( Site 2603), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University-Oncology ( Site 2607), Xi'an, Shaanxi
  - Shandong Cancer Hospital-Oncology Department ( Site 2630), Jinan, Shandong
  - Fudan University Shanghai Cancer Center ( Site 2616), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital-Oncology Department ( Site 2601), Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital ( Site 2628), Chengdu, Sichuan
  - West China Hospital of Sichuan University ( Site 2610), Chengdu, Sichuan
  - The Second People's Hospital of Yibin ( Site 2629), Yibin, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital-lung cancer ( Site 2606), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University-Respiratory Department ( Site 2613), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 2615), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Oncology ( Site 2612), Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine-Respiratory Medicine ( Site, Hangzhou, Zhejiang
- Colombia (5):
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 0603), Medellín, Antioquia
  - Administradora Country S.A. - Clinica del Country ( Site 0601), Bogotá, Bogota D.C.
  - Sociedad De Oncologia Y Hematologia Del Cesar ( Site 0606), Valledupar, Cesar Department
  - Oncomedica S.A.-Oncomedica S.A ( Site 0609), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 0608), Pereira, Risaralda Department
- France (7):
  - CENTRE HOSPITALIER REGIONAL D'ORLEANS-Service de Pneumologie ( Site 0806), Orléans, Centre-Val de Loire
  - Centre Hospitalier d'Annecy ( Site 0807), Epagny Metz-Tessy, Haute-Savoie
  - Centre Hospitalier Regional Universitaire de Lille - Hôpital-Service de pneumologie et oncologie th, Lille, Hauts-de-France
  - Institut de Cancérologie de l'Ouest ( Site 0802), Angers, Maine-et-Loire
  - CENTRE LEON BERARD ( Site 0803), Lyon, Rhone
  - HIA Sainte Anne ( Site 0804), Toulon, Var
  - Centre Hospitalier d'Avignon ( Site 0810), Avignon, Vaucluse
- Germany (5):
  - UKGM Gießen/Marburg-Medical Clinic V ( Site 0912), Giessen, Hesse
  - GEFOS Gesellschaft f. onkologische Studien ( Site 0909), Dortmund, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein-Pneumologie ( Site 0902), Lübeck, Schleswig-Holstein
  - SRH Wald-Klinikum Gera ( Site 0911), Gera, Thuringia
  - Charité Campus Virchow-Klinikum-Department of Infectious Diseases and Pulmonary Medicine ( Site 0913, Berlin
- Israel (5):
  - Rambam Health Care Campus-Oncology ( Site 1303), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 1306), Jerusalem
  - Meir Medical Center-oncology ( Site 1301), Kfar Saba
  - Sheba Medical Center-ONCOLOGY ( Site 1302), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 1305), Tel Aviv
- Japan (15):
  - National Hospital Organization Shikoku Cancer Center ( Site 2414), Matsuyama, Ehime
  - Ehime University Hospital ( Site 2411), Tōon, Ehime
  - Hyogo Cancer Center-Thoracic Oncology ( Site 2409), Akashi, Hyōgo
  - Kanazawa University Hospital ( Site 2407), Kanazawa, Ishikawa-ken
  - Kanagawa cancer center-Department of Thoracic Oncology ( Site 2405), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 2401), Natori-shi, Miyagi
  - Kansai Medical University Hospital ( Site 2415), Hirakata, Osaka
  - Saitama Prefectural Cancer Center ( Site 2406), Ina-machi, Saitama
  - Shizuoka Cancer Center ( Site 2408), Nakatogari, Shizuoka
  - Japanese Foundation for Cancer Research ( Site 2402), Koto, Tokyo
  - Showa University Hospital ( Site 2403), Shinagawa, Tokyo
  - National Hospital Organization Kyushu Medical Center ( Site 2413), Fukuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 2412), Fukuoka
  - Okayama University Hospital ( Site 2410), Okayama
  - Nippon Medical School Hospital ( Site 2404), Tokyo
- Mexico (4):
  - CENTRO DE INFUSION E INVESTIGACION ONCOLOGIA DE SALTILLO S.C. ( Site 0304), Saltillo, Coahuila
  - Hospital Civil Fray Antonio Alcalde ( Site 0307), Guadalajara, Jalisco
  - Arké SMO S.A. de C.V. ( Site 0301), Mexico City, Mexico City
  - Alivia Clínica de Alta Especialidad ( Site 0310), Mexico City, Mexico City
- Poland (8):
  - Przychodnia Lekarska KOMED ( Site 1902), Konin, Greater Poland Voivodeship
  - Med-Polonia Sp. z o. o. ( Site 1909), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1903), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Ostrobramska NZOZ Magodent ( Site 1908), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1904), Przemyśl, Podkarpackie Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o. ( Site 1906), Prabuty, Pomeranian Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej ( Site 1907), Bystra, Silesian Voivodeship
- South Korea (6):
  - Chonnam National University Hwasun Hospital-Pulmonology ( Site 2201), Hwasun, Jeonranamdo
  - Pusan National University Hospital ( Site 2205), Busan, Pusan-Kwangyokshi
  - Asan Medical Center ( Site 2206), Songpa-gu, Seoul
  - Kyungpook National University Chilgok Hospital-Pulmonology ( Site 2202), Deagu, Taegu-Kwangyokshi
  - Chungnam national university hospital-Department of Internal Medicine ( Site 2203), Daejeon, Taejon-Kwangyokshi
  - Korea University Guro Hospital-Internal Medicine ( Site 2204), Seoul
- Spain (6):
  - CHUAC-Hospital Teresa Herrera-MEDICAL ONCOLOGY ( Site 1106), A Coruña, La Coruna
  - Hospital Insular de Gran Canaria-Oncology ( Site 1102), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1101), Barcelona
  - Hospital Clinico San Carlos-Oncology Department ( Site 1107), Madrid
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 1103), Seville
  - Hospital Clínico Universitario Lozano Blesa-Oncology ( Site 1105), Zaragoza
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 2254), Kaohsiung City
  - China Medical University Hospital ( Site 2253), Taichung
  - NATIONAL CHENG-KUNG UNI. HOSP. ( Site 2252), Tainan
  - National Taiwan University Hospital-Oncology ( Site 2255), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 2251), Taoyuan District
- Thailand (5):
  - Faculty of Medicine Siriraj Hospital ( Site 2304), Bangkok, Bangkok
  - Chulabhorn Hospital ( Site 2305), Lak Si, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 2303), Muang, Changwat Khon Kaen
  - Songklanagarind hospital ( Site 2302), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital-Chiang Mai Clinical Trial Unit (CM-CTU) ( Site 2301), Chiang Mai
- Turkey (Türkiye) (8):
  - Acibadem Altunizade Hospital-Oncology ( Site 1207), Üsküdar / Stanbul, Istanbul
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 1208), Adana
  - Hacettepe Universitesi-oncology hospital ( Site 1202), Ankara
  - Liv Hospital Ankara-Oncology ( Site 1205), Ankara
  - Ankara City Hospital ( Site 1204), Ankara
  - Trakya University-Medical Oncology ( Site 1203), Edirne
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1209), Istanbul
  - Umraniye Training and Research Hospital-medical oncology ( Site 1206), Istanbul
- United Kingdom (4):
  - Leicester Royal Infirmary-HOPE Clinical Trials Unit ( Site 1502), Leicester, England
  - Chelsea and Westminster Hospital NHS Foundation Trust-Research and Development ( Site 1501), London, England
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 1506), London, London, City of
  - University College London Hospital-Cancer Clinical Trials Unit ( Site 1509), London-Camden, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Shapira-Frommer R, Niu J, Perets R, Peters S, Shouse G, Lugowska I, Garassino MC, Sands J, Keenan T, Zhao B, Healy J, Ahn MJ. The KEYVIBE program: vibostolimab and pembrolizumab for the treatment of advanced malignancies. Future Oncol. 2024;20(27):1983-1991. doi: 10.1080/14796694.2024.2343272. Epub 2024 Sep 4. PMID 39230120
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26241&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-7684A + Chemotherapy: Participants receive MK-7684A (co-formulation of 200mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 35 cycles (up to ~2 years) PLUS paclitaxel IV (on Day 1 of each cycle) OR nab-paclitaxel IV (on Days 1, 8, and 15 of each cycle) and carboplatin IV (on Day 1 of each cycle) for 4 cycles for Squamous non-small cell lung cancer (NSCLC); PLUS carboplatin IV (on Day 1 of each cycle) or cisplatin IV (on Day 1 of each cycle) for 4 cycles and pemetrexed IV (on Day 1 of each cycle) until progression, intolerable adverse events, or participant/physician decision for Non-squamous.
Period: Overall Study
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Started | 366 | 373
Treated | 360 | 368
Transitioned to Pembrolizumab + Chemotherapy | 0 | 0
Completed | 0 | 0
Not Completed | 366 | 373
Not completed — Death | 186 | 191
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Ongoing | 174 | 176

BASELINE CHARACTERISTICS:
Groups:
- MK-7684A + Chemotherapy: Participants receive MK-7684A (co-formulation of 200mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 35 cycles (up to ~2 years) PLUS paclitaxel IV (on Day 1 of each cycle) OR nab-paclitaxel IV (on Days 1, 8, and 15 of each cycle) and carboplatin IV (on Day 1 of each cycle) for 4 cycles for Squamous NSCLC; PLUS carboplatin IV (on Day 1 of each cycle) or cisplatin IV (on Day 1 of each cycle) for 4 cycles and pemetrexed IV (on Day 1 of each cycle) until progression, intolerable adverse events, or participant/physician decision for Non-squamous.
- Total: Total of all reporting groups
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy | Total
Number analyzed (Participants) | 366 | 373 | 739
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.3) | 64.3 (8.9) | 64.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 121 | 219
  Male | 268 | 252 | 520
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98 | 92 | 190
  Not Hispanic or Latino | 231 | 249 | 480
  Unknown or Not Reported | 37 | 32 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 22 | 50
  Asian | 125 | 131 | 256
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 196 | 210 | 406
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Programmed Cell Death-Ligand 1 (PD-L1) Tumor Proportion Score (TPS) ≥1%
Description: OS is defined as the time from the date of randomization to death due to any cause. The OS is reported for all participants with PD-L1 positive tumors (PD-L1 TPS≥1%). The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: The analysis population includes all randomized participants with PD-L1 TPS≥1%. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 240 | 213
Months | 19.4 [17.2 to 23.9] | 23.5 [19.6 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: MK-7684A + Chemotherapy vs Pembrolizumab + Chemotherapy; Test type: Superiority; p = 0.8335, Log Rank — One-sided p-value based on log-rank test stratified by ECOG, predominant tumor histology, PD-L1 expression, and geographic region; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.87 to 1.50] — Based on Cox regression model with Efron's method of tie handling; treatment as covariate stratified by ECOG, predominant tumor histology, PD-L1 expression, and geographic region

2. Secondary Outcome: Overall Survival (OS) in All Participants
Description: OS is defined as the time from the date of randomization to death due to any cause. The OS is reported for all randomized participants. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: The analysis population includes all randomized participants. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 366 | 373
Months | 20.0 [17.0 to 22.5] | 19.7 [17.5 to 23.4]
Statistical Analysis 1: Comparison: MK-7684A + Chemotherapy vs Pembrolizumab + Chemotherapy; Test type: Superiority; p = 0.5104, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.82 to 1.23] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) was planned to be presented.
Time Frame: Up to approximately 29 months
Population: After additional Futility Analysis of OS was performed before the first efficacy analysis, as per the supplemental Statistical Analysis Plan amendment (effective date: September 16, 2025) it was stated that no further efficacy analyses would be performed, so the originally planned PFS data are unavailable.
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by blinded independent central review (BICR) was planned to be presented.
Time Frame: Up to approximately 29 months
Population: After additional Futility Analysis of OS was performed before the first efficacy analysis, as per the supplemental Statistical Analysis Plan amendment (effective date: September 16, 2025) it was stated that no further efficacy analyses would be performed, so the originally planned ORR data are unavailable.
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrate a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by BICR was planned to be presented.
Time Frame: Up to approximately 29 months
Population: After additional Futility Analysis of OS was performed before the first efficacy analysis, as per the supplemental Statistical Analysis Plan amendment (effective date: September 16, 2025) it was stated that no further efficacy analyses would be performed, so the originally planned DOR data are unavailable.
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
Description: Change from baseline in the score of EORTC QLQ-C30 Items 29 and 30 was planned to be presented. The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome.
Time Frame: Baseline and Up to approximately 29 months
Population: After additional Futility Analysis of OS was performed before the first efficacy analysis, as per the supplemental Statistical Analysis Plan amendment (effective date: September 16, 2025) it was stated that no further efficacy analyses would be performed, so the originally planned electronic patient-reported outcome (ePRO) data are unavailable.
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30
Description: Change from baseline in the score of EORTC QLQ-C30 Items 1-5 was planned to be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function.
Time Frame: Baseline and Up to approximately 29 months
Population: After additional Futility Analysis of OS was performed before the first efficacy analysis, as per the supplemental Statistical Analysis Plan amendment (effective date: September 16, 2025) it was stated that no further efficacy analyses would be performed, so the originally planned ePRO data are unavailable.
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline for Role Functioning (Items 6 and 7) Combined Score on the EORTC QLQ-C30
Description: Change from baseline in the score of EORTC QLQ-C30 Items 6-7 was planned to be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function.
Time Frame: Baseline and up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30
Description: Change from baseline in the score of EORTC QLQ-C30 Item 8 was planned to be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea.
Time Frame: Baseline and Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Cough Score (Item 31) on the European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire Module (EORTC QLQ-LC13)
Description: Change from baseline in the score of EORTC QLQ-LC13 Item 31 was planned to be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing.
Time Frame: Baseline and Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Chest Pain Score (Item 40) on the EORTC QLQ- LC13
Description: Change from baseline in the score of EORTC QLQ-LC13 Item 40 was planned to be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain.
Time Frame: Baseline and Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Time to Deterioration (TTD) in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the EORTC QLQ-C30
Description: TTD in the score of EORTC QLQ-C30 Items 29 and 30 was planned to be presented. The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ- C30
Description: TTD in the score of EORTC QLQ-C30 Items 1-5 was planned to be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: TTD in Role Functioning (Items 6 and 7) Combined Score on the EORTC QLQ-C30
Description: TTD in the score of EORTC QLQ-C30 Items 6-7 was planned to be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30
Description: TTD in the score of EORTC QLQ-C30 Item 8 was planned to be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: TTD in Cough Score (Item 31) on the EORTC QLQ-LC13
Description: TTD in the score of EORTC QLQ-LC13 Item 31 was planned to be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: TTD in Chest Pain Score (Item 40) on the EORTC QLQ-LC13
Description: TTD in the score of EORTC QLQ-LC13 Item 40 was planned to be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Up to approximately 29 months
Population: as for outcome 7
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: The number of participants who experienced an adverse event (AE) will be presented. An AE is defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to approximately 46 months
Reporting Status: Not Posted, anticipated posting 2027-01

19. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: The number of participants who discontinue study intervention due to an adverse event (AE) will be presented. An AE is defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to approximately 46 months
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Time Frame: Up to approximately 29 months
Description: The population for all-cause mortality includes all participants. AE populations include all randomized participants who received at least 1 dose of study drug. Terms 'Neoplasm progression' 'Malignant neoplasm progression' and 'Disease progression' not related to the drug are excluded.
Arm/Group | MK-7684A + Chemotherapy | Pembrolizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 190/366 | 193/373
Serious Adverse Events (participants affected / at risk) | 205/360 | 180/368
Other Adverse Events (participants affected / at risk) | 349/360 | 352/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7684A + Chemotherapy (N=360) | Pembrolizumab + Chemotherapy (N=368)
Anaemia (Blood and lymphatic system disorders) | 16 (18) | 15 (17)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 5 (7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 3 (3)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 7 (7)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (3)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 4 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 3 (3) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 2 (2)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (2) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 6 (6)
Fatigue (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (2)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Inadequate analgesia (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 4 (4)
Treatment noncompliance (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 1 (1) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clonorchiasis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Myiasis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 42 (50) | 38 (49)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia fungal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 10 (10) | 5 (5)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (8) | 6 (6)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (7) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 12 (12)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7684A + Chemotherapy (N=360) | Pembrolizumab + Chemotherapy (N=368)
Anaemia (Blood and lymphatic system disorders) | 228 (392) | 231 (368)
Neutropenia (Blood and lymphatic system disorders) | 143 (303) | 125 (319)
Thrombocytopenia (Blood and lymphatic system disorders) | 102 (173) | 101 (176)
Hyperthyroidism (Endocrine disorders) | 24 (24) | 21 (23)
Hypothyroidism (Endocrine disorders) | 50 (59) | 44 (53)
Constipation (Gastrointestinal disorders) | 91 (112) | 95 (105)
Diarrhoea (Gastrointestinal disorders) | 75 (95) | 57 (89)
Nausea (Gastrointestinal disorders) | 121 (208) | 117 (216)
Vomiting (Gastrointestinal disorders) | 57 (89) | 40 (51)
Asthenia (General disorders) | 79 (109) | 80 (128)
Chest pain (General disorders) | 15 (20) | 29 (37)
Fatigue (General disorders) | 78 (116) | 71 (100)
Oedema peripheral (General disorders) | 47 (59) | 43 (52)
Pyrexia (General disorders) | 32 (43) | 34 (43)
COVID-19 (Infections and infestations) | 36 (37) | 30 (32)
Nasopharyngitis (Infections and infestations) | 13 (21) | 20 (27)
Pneumonia (Infections and infestations) | 24 (24) | 23 (32)
Urinary tract infection (Infections and infestations) | 21 (22) | 30 (41)
Alanine aminotransferase increased (Investigations) | 93 (155) | 94 (143)
Amylase increased (Investigations) | 60 (106) | 38 (64)
Aspartate aminotransferase increased (Investigations) | 87 (140) | 90 (169)
Blood alkaline phosphatase increased (Investigations) | 35 (57) | 37 (58)
Blood creatinine increased (Investigations) | 59 (103) | 55 (76)
Blood lactate dehydrogenase increased (Investigations) | 36 (60) | 36 (56)
Gamma-glutamyltransferase increased (Investigations) | 29 (37) | 39 (56)
Lipase increased (Investigations) | 45 (86) | 42 (68)
Lymphocyte count decreased (Investigations) | 51 (109) | 32 (69)
Weight decreased (Investigations) | 64 (74) | 50 (57)
Weight increased (Investigations) | 26 (27) | 13 (14)
White blood cell count decreased (Investigations) | 100 (269) | 88 (215)
Decreased appetite (Metabolism and nutrition disorders) | 91 (132) | 75 (103)
Hyperglycaemia (Metabolism and nutrition disorders) | 37 (55) | 37 (65)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 49 (80) | 59 (107)
Hypocalcaemia (Metabolism and nutrition disorders) | 29 (40) | 19 (28)
Hypokalaemia (Metabolism and nutrition disorders) | 41 (57) | 38 (55)
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 (53) | 32 (50)
Hyponatraemia (Metabolism and nutrition disorders) | 41 (60) | 39 (59)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (53) | 40 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (35) | 20 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 24 (29) | 26 (44)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (32) | 29 (38)
Dizziness (Nervous system disorders) | 25 (34) | 23 (31)
Headache (Nervous system disorders) | 22 (23) | 28 (52)
Neuropathy peripheral (Nervous system disorders) | 25 (27) | 34 (41)
Insomnia (Psychiatric disorders) | 43 (48) | 29 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 61 (69) | 40 (49)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 37 (43)
Alopecia (Skin and subcutaneous tissue disorders) | 55 (55) | 39 (39)
Pruritus (Skin and subcutaneous tissue disorders) | 107 (149) | 50 (62)
Rash (Skin and subcutaneous tissue disorders) | 95 (149) | 55 (72)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 24 (43) | 13 (17)

LIMITATIONS AND CAVEATS:
The pre-specified futility criteria were met at the futility analysis before efficacy IA, and the Sponsor decided to discontinue treatment with MK 7684A. No additional efficacy analysis will be conducted. Analyses on secondary efficacy endpoints, specifically PFS, ORR, DOR and patient-reported outcomes (PROs), will not be conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT05226598/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT05226598/SAP_001.pdf